CLINICAL TRIAL: NCT01582282
Title: A Clinical Study to Determine the Ability of Metamucil to Reduce Fasting Blood Glucose and HbA1c Levels in Type II NIDDM
Brief Title: Study of Metamucil on Blood Glucose and HbA1c in Type II NIDDM Subjects
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: due to slow enrollment
Sponsor: Procter and Gamble (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: LX-105
Record Dates: First submitted 2012-04-18; First posted 2012-04-20 (Estimated); Results first posted 2012-11-02 (Estimated); Last update posted 2012-11-15 (Estimated); Status verified 2012-11

CONDITIONS: Non-Insulin-dependent Diabetes Mellitus
Keywords: Type II NIDDM
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Psyllium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- placebo (Placebo Comparator): matched placebo BID
  Interventions: Dietary Supplement: placebo
- psyllium 3.4g BID (Active Comparator): 3.4g psyllium BID for a Total of 6.8g daily
  Interventions: Dietary Supplement: 3.4 g psyllium BID
- 6.8g psyllium BID (Active Comparator): 6.8g psyllium BID for a total of 13.6 g/day
  Interventions: Dietary Supplement: 6.8g psyllium BID

INTERVENTIONS:
Dietary Supplement: placebo — fiber-free placebo
  Arms: placebo
Dietary Supplement: 3.4 g psyllium BID — 3.4 g psyllium BID for a total of 6.8 g/day (10.4g Metamucil)
  Other Names: Metamucil
  Arms: psyllium 3.4g BID
Dietary Supplement: 6.8g psyllium BID — 6.8g psyllium BID for a total of 13.6 g/day (20.8g Metamucil)
  Other Names: Metamucil
  Arms: 6.8g psyllium BID

SUMMARY:
A double-blind, randomized, placebo-controlled, multi-dose clinical study consisting of 2 phases; 1) an 8-week lead-in period during which patients followed a diet judged to be within the acceptable guidelines of the ADA, and 2) a 12-week treatment period, at the beginning of which, Subjects are randomly assigned to 1 of the 3 treatment groups: placebo, 3.4 g psyllium BID for a total of 6.8 g/day (10.4g Metamucil) or 6.8g psyllium BID for a total of 13.6 g/day (20.8g Metamucil). For 12 weeks, Subjects took Metamucil or the fiber-free placebo BID, just prior to breakfast and dinner.

Patients visited the clinic 10 times during the 20-week period at Screening, Weeks -8, -6, -4, 0, Day 3, and Weeks 2, 4, 8 and 12, fasting at least 12 hours prior to each visit where a blood sample was taken (all visits except Week -6 and Day 3) for analysis of fasting serum glucose and lipid levels, and HbA1c. Clinical chemistry, hematology and urinalysis were done at Weeks -8, 0 and 12. The completed 7-day food diaries were reviewed by the study dietician at each visit and discussed with the patient to ensure compliance with the recommended diet and the patients' body weights were recorded

DETAILED DESCRIPTION:
During the first phase, lead-in period during Subjects followed a diet judged to be within the acceptable guidelines of the ADA, with compliance assessed by a study dietician using 7-day food diaries completed by the patients. Subject body weight, serum glucose and serum HbA1c, and lipid levels were allowed to stabilize during this period.

During the 12-week treatment period, Subjects were stratified by either diet alone or diet and oral hypoglycemic medication and randomly assigned to 1 of the 3 treatment groups: placebo, 3.4 g psyllium BID for a total of 6.8 g/day (10.4g Metamucil) or 6.8g psyllium BID for a total of 13.6 g/day (20.8g Metamucil). For 12 weeks, patients took Metamucil or the fiber-free placebo BID, just prior to breakfast and dinner.

Patients visited the clinic 10 times during the 20-week period at Screening, Weeks -8, -6, -4, 0, Day 3, and Weeks 2, 4, 8 and 12, fasting at least 12 hours prior to each visit where a blood sample was taken (all visits except Week -6 and Day 3) for analysis of fasting serum glucose and lipid levels, and HbA1c. Clinical chemistry, hematology and urinalysis were done at Weeks -8, 0 and 12. The completed 7-day food diaries were reviewed by the study dietician at each visit and discussed with the patient to ensure compliance with the recommended diet and the patients' body weights were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Have a clinical diagnosis of Type II diabetes mellitus, controlled by diet and/or second generation oral hypoglycemic drugs, with the onset of the disease after age 35.
* Are between 0 and 50% above "normal" body weight (adjusted by frame) according to the Metropolitan Life Insurance Tables.
* Are male or female, aged 36-80 years with a diagnosis made at least 1 year prior to enrollment.
* Have an HbA1c level between 6 and 10%
* Have a fasting serum glucose level between 120-220 mg/dL and not vary by more than ±20% during the month prior to entering the treatment phase and HbA1c levels not vary by more than ±10% during the month prior to entering the treatment phase. Serum glucose level must have been between 120-220mg/dl and the subject's HbA1c between 6 and 10% at Week 0.
* Have been on a "stable" diet consistent with ADA-recommended dietary guidelines with intake of total dietary fiber < 15g/1000 calories and were willing to maintain this diet during the 20-week study.
* Have maintained a constant body weight (±5%) during the month prior to entering the treatment phase

Exclusion Criteria:

* Have a condition that would interfere with evaluation

Ages: 36 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 1988-05; Primary Completion 1990-01 (Actual); Study Completion 1990-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Reeves, MD, Principal Investigator — University of Miami; Richard Bergenstal, MD, Principal Investigator — International Diabetes Center, Minneapolis, MN 55416
Locations (2):
- United States (2):
  - University of Miami, Diabetes Unit D-1, Miami, Florida
  - International Diabetes Center, Minneapolis, Minnesota

RESULTS

PARTICIPANT FLOW:
Groups:
- Psyllium 3.4g BID: Metamucil, psyllium 3.4g BID (6.8g/day)
- 6.8g Psyllium BID: Metamucil, psyllium 6.8g BID (13.6g/day)
- Placebo: Placebo, orange-flavored formulation with excipients of the Metamucil formulation without psyllium BID
Period: Overall Study
Arm/Group | Psyllium 3.4g BID | 6.8g Psyllium BID | Placebo
Started | 15 | 14 | 8
Completed | 13 | 12 | 8
Not Completed | 2 | 2 | 0
Not completed — Adverse Event | 1 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — fasting blood glucose outside Protocol | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Psyllium 3.4g BID | 6.8g Psyllium BID | Placebo | Total
Number analyzed (Participants) | 15 | 14 | 8 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 15 | 14 | 8 | 37
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 61.8 (9.39) | 64.8 (8.42) | 56.5 (9.99) | 61.8 (9.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 2 | 12
  Male | 10 | 9 | 6 | 25
Region of Enrollment [Number; unit: participants]
  United States | 15 | 14 | 8 | 37

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Fasting Glucose
Description: Change from Baseline is defined as the Post-Baseline value subtracted from the Baseline value
Time Frame: 12 weeks
Population: Intent-to-Treat
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Psyllium 3.4g BID | 6.8g Psyllium BID | Placebo
Number analyzed (Participants) | 13 | 12 | 8
mg/dL | -7.73 (8.02) | -17.81 (8.81) | 22.91 (10.71)
Statistical Analysis 1: Comparison: Psyllium 3.4g BID vs Placebo; Test type: Superiority or Other; p = 0.028, ANCOVA; Mean Difference (Final Values) = 30.64
Statistical Analysis 2: Comparison: 6.8g Psyllium BID vs Placebo; Test type: Superiority or Other; p = 0.009, ANCOVA; Mean Difference (Final Values) = 40.72

2. Primary Outcome: Change From Baseline in Fasting HbA1c
Description: Change is defined as Post-Baseline minus Baseline
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: percentage of total hemoglobin
Arm/Group | Psyllium 3.4g BID | 6.8g Psyllium BID | Placebo
Number analyzed (Participants) | 13 | 12 | 8
percentage of total hemoglobin | -0.27 (0.12) | -0.39 (0.13) | 0.26 (0.16)
Statistical Analysis 1: Comparison: Psyllium 3.4g BID vs Placebo; Test type: Superiority or Other; p = 0.013, ANCOVA; Mean Difference (Final Values) = 0.53
Statistical Analysis 2: Comparison: 6.8g Psyllium BID vs Placebo; Test type: Superiority or Other; p = 0.003, ANCOVA; Mean Difference (Final Values) = 0.65

3. Primary Outcome: Change From Baseline in Fasting HDL Cholesterol
Description: Change is defined as Post-Baseline minus Baseline
Time Frame: 12 weeks
Population: Analysis of Covariance of Cholesterol Measures Intent-to-Treat
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Psyllium 3.4g BID | 6.8g Psyllium BID | Placebo
Number analyzed (Participants) | 13 | 12 | 8
mg/dL | -0.90 (1.21) | 1.58 (1.27) | -0.42 (1.54)
Statistical Analysis 1: Comparison: Psyllium 3.4g BID vs Placebo; Test type: Superiority or Other; p = 0.808, ANCOVA; Mean Difference (Final Values) = 0.48
Statistical Analysis 2: Comparison: 6.8g Psyllium BID vs Placebo; Test type: Superiority or Other; p = 0.328, ANCOVA; Mean Difference (Final Values) = -2.0

4. Primary Outcome: Change From Baseline in Fasting LDL Cholesterol
Description: Change is defined as Post-Baseline minus Baseline
Time Frame: 12 weeks
Population: The LDL cholesterol values for two subjects at week 12 were unreportable.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Psyllium 3.4g BID | 6.8g Psyllium BID | Placebo
Number analyzed (Participants) | 11 | 12 | 8
mg/dL | -11.51 (5.86) | -5.84 (5.59) | -5.41 (6.89)
Statistical Analysis 1: Comparison: Psyllium 3.4g BID vs Placebo; Test type: Superiority or Other; p = 0.508, ANCOVA; Mean Difference (Final Values) = 6.1
Statistical Analysis 2: Comparison: 6.8g Psyllium BID vs Placebo; Test type: Superiority or Other; p = 0.962, ANCOVA; Mean Difference (Final Values) = 0.43

5. Primary Outcome: Total Cholesterol Change From Baseline
Description: Change is defined as Post-Baseline minus Baseline
Time Frame: 12 weeks
Population: Analysis of Covariance of Cholesterol Measures Intent-to-Treat
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Psyllium 3.4g BID | 6.8g Psyllium BID | Placebo
Number analyzed (Participants) | 13 | 12 | 8
mg/dL | -12.96 (5.22) | -4.88 (5.43) | -5.12 (6.66)
Statistical Analysis 1: Comparison: Psyllium 3.4g BID vs Placebo; Test type: Superiority or Other; p = 0.363, ANCOVA; Mean Difference (Final Values) = 7.84
Statistical Analysis 2: Comparison: 6.8g Psyllium BID vs Placebo; Test type: Superiority or Other; p = 0.978, ANCOVA; Mean Difference (Final Values) = -.24

6. Primary Outcome: Triglyceride Change From Baseline
Description: Change is defined as Post-Baseline minus Baseline
Time Frame: 12 weeks
Population: Analysis of Covariance of Cholesterol Measures Intent-to-Treat
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Psyllium 3.4g BID | 6.8g Psyllium BID | Placebo
Number analyzed (Participants) | 13 | 12 | 8
mg/dL | -8.95 (16.22) | -8.26 (17.03) | -1.81 (20.41)
Statistical Analysis 1: Comparison: Psyllium 3.4g BID vs Placebo; Test type: Superiority or Other; p = 0.785, ANCOVA; Mean Difference (Final Values) = 7.14
Statistical Analysis 2: Comparison: 6.8g Psyllium BID vs Placebo; Test type: Superiority or Other; p = 0.811, ANCOVA; Mean Difference (Final Values) = 6.45

ADVERSE EVENTS:
Time Frame: through 12 weeks
Arm/Group | Psyllium 3.4g BID | 6.8g Psyllium BID | Placebo
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/14 | 0/8
Other Adverse Events (participants affected / at risk) | 12/15 | 12/14 | 7/8
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Psyllium 3.4g BID (N=15) | 6.8g Psyllium BID (N=14) | Placebo (N=8)
Abdominal Discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abnormal faeces (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 4 (4) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Faecal volume increased (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 5 (6) | 5 (6) | 1 (1)
Frequent bowel movements (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Stools abnormal (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Stool analysis abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Nervousness (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Data, calculations, interpretations, opinions, and recommendations are the property of P&GP